CLINICAL TRIAL: NCT00754078
Title: A Phase II Study to Assess Acute Toxicity and Quality of Life of Patients With Carcinoma of the Anal Canal Receiving Chemotherapy and Radiation Using Helical Tomotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GI-24329
Record Dates: First submitted 2008-09-15; First posted 2008-09-17 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Anal Canal Cancer
Keywords: tomotherapy
MeSH Terms: conditions — Anal Canal Carcinoma | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): anal cancer patients treated with tomotherapy and chemotherapy
  Interventions: Radiation: Tomotherapy

INTERVENTIONS:
Radiation: Tomotherapy — 30 fractions of tomotherapy treatment

SUMMARY:
The hypothesis is that helical tomotherapy could minimize radiation related toxicity by avoiding or limiting doses to structures such as small bowel, external genitalia, skin, bladder, rectum, and femoral neck and head.

DETAILED DESCRIPTION:
This is a phase II study using tomotherapy for radiation treatment delivery along with concurrent 5-FU/mitomycin C for the treatment of T2-T4 cancer of the anal canal. They hypothesis is that helical tomotherapy could minimize radiation related toxicity by avoiding or limiting doses to structures such as small bowel, external genitalia, skin, bladder, rectum, and femoral neck and head. This is expected to limit or reduce treatment related toxicity and hence prevent or reduce treatment breaks. This may result in delivery of radical treatment with better local control and treatment outcome than using the current radiation treatment technique at our center.

ELIGIBILITY:
Inclusion Criteria:

* Patient should have histologically proven primary squamous carcinoma or its variant
* No history of prior malignancy.
* Patients must be free of metastatic disease out of pelvis at the time of diagnosis
* Patients must be at least 18 years of age
* Performance status 0, 1 or 2 ECOG
* T stage 2-4, Any N, stage MO
* Patient should be eligible for concomitant chemotherapy
* Informed written consent required to participate

Exclusion Criteria:

* Prior radiation to pelvis
* Pregnant or lactating
* prior surgical treatment for anal cancer other than biopsy
* prior surgical or chemotherapy treatment for anal cancer
* T1 tumours (2cm) or evidence of distant mets
* comorbid medical conditions precluding radical treatment at the discretion of oncologist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2008-09; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Acute Toxicity and Quality of LIfe | 3 months

SECONDARY OUTCOMES:
colostomy-free survival and/or overall survival | 3 and 5 years
Local Recurrence | 3 and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Kurian J Joseph, MD, FRCPC, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada